CLINICAL TRIAL: NCT03324074
Title: Assessment of Pyloric Sphincter Physiology Using EndoFLIP
Brief Title: Assessment of Pyloric Sphincter Physiology
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh K, Principal Investigator, Asian Institute of Gastroenterology, India
Other Study IDs: EndoFLIP01.Ver.01.
Record Dates: First submitted 2017-10-17; First posted 2017-10-27 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Physiology of Pyloric Sphincter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pylorus is a tubular structure which contains circular muscle, forming pyloric sphincter which separates stomach and duodenum. The motor activity of the pyloric sphincter is less investigated. Antroduodenal manometry is an invasive and time consuming technique also limited by inability to measure compliance of the sphincter.

Recently, a new technique functional lumen imaging probe (FLIP) which is based on principle of impedance planimetry (IP). The endoluminal FLIP (EndoFLIP) EF -100 system uses a multi-detector IP system to produce a 3-dimensional outline of a sphincter. EndoFLIP can measure tissue distensibility and geometric changes through volumetric distention with real-time images. The esophagogastric junction (EGJ) has been well studied using EndoFLIP, studies for assessment of pyloric function are lacking.

DETAILED DESCRIPTION:
Objective:

To evaluate the motor activity of pyloric sphincter using Endo FLIP in the form of pressure, diameter, cross-sectional area (CSA) and distensibility in the healthy volunteers.

Methods 20 healthy volunteers will be recruited by local advertising, hospital staff and hospitalised patient's relatives. They will be screened for evidence of organic or functional gastrointestinal disorders, if found to have any will be excluded. Subjects on any medication that is known to affect gastrointestinal function will be excluded.

EndoFLIP method

The subjects will be fasting for at least 8 hours prior to the study. The study will be performed under sedation using monitored anesthesia using propofol in the left lateral decubitus position. Initial endoscopic examination will be performed up to the antrum without traversing the pylorus using (160 Olympus).An EndoFLIP catheter will be passed through biopsy channel into pylorus under direct endoscopic and fluoroscopic visualization.

Pylorus will be assessed using EndoFLIP at 20, 30, 40 and 50 cc balloon volume distentions. Pressure will be measured by pressure transducer inside the balloon. CSA will be measured using impedance planimetry by Ohm's Law. Distensibility will be calculated as minimum CSA divided by pressure at each balloon fill volume. These measurement will be assessed after the balloon inflated at each balloon distension for minimum of 5 seconds. The length of the pylorus will be assessed visually from EndoFLIP images. Once the EndoFLIP measurements completed at rest, Injection hyoscine 10mg intravascular will be administered, and same measurements will be repeated. Thereafter remaining endoscopic exam will be completed.

This is an observational study with no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years and < 60 years, Both males and females.
* Healthy volunteers willing to give written informed consent.

Exclusion Criteria:

* Patient younger than 18 years or older than 80 years
* Pregnancy or breast feeding
* Previous history of esophago-gastric surgery or vagotomy
* Previous history of Parkinson disease or diabetes mellitus
* Contra-indication to upper gastro-intestinal endoscopy
* Esophageal varices
* Esophageal diameter smaller than 5 mm
* Contra-indication to general anesthesia
* Hiatal hernia greater than 3 cm on endoscopy
* Esophageal or gastric cancer otherwise than superficial lesion with indication of submucosal dissection
* Typical symptoms (heartburn, regurgitation) of gastro-esophageal reflux disease and/or gastroesophageal reflux disease (GERD)-Q score greater or equal to 8
* Nausea, vomiting or epigastric pain
* Dysphagia with Sydney score greater or equal to 50
* Incapability to give consent
* No written informed consent
* Participation to another study at the same time

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion Criteria:
  * Adult >18 years and < 60 years, Both males and females.
  * Healthy volunteers willing to give written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Assessment of pyloric sphincter pressure | 1 day
  To evaluate the pyloric sphincter pressure using EndoFLIP in the healthy volunteers.
Assessment of pyloric sphincter diameter | 1 day
  To evaluate the pyloric sphincter diameter using EndoFLIP in the healthy volunteers.
Assessment of pyloric sphincter cross-sectional area | 1 day
  To evaluate the pyloric sphincter cross-sectional area using EndoFLIP in the healthy volunteers.
Assessment of pyloric sphincter distensibility | 1 day
  To evaluate the pyloric sphincter distensibility using EndoFLIP in the healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. D. Nageshwar Reddy, MD,DM, Study Director — Asian Institute of Gastroenterology
Locations (1):
- Rakesh K, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No